CLINICAL TRIAL: NCT03884647
Title: DELPHI Software for the Analysis of TMS-EEG Data of Brain Functionality - in Subjects at Risk for Stroke and Dementia
Brief Title: DELPHI in Subjects at Risk for Stroke and Dementia
Status: Completed | Type: Observational
Sponsor: QuantalX Neuroscience (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-10-410
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-02

CONDITIONS: Stroke; Hypertension; Diabete Mellitus; Dyslipidemias; Sleep Disorder; Smoking; Overweight and Obesity; Familial Alzheimer Disease; Atrial Fibrillation; Cardiac Disease; Cognitive Impairment; Transient Ischemic Attack
MeSH Terms: conditions — Stroke; Hypertension; Diabetes Mellitus; Dyslipidemias; Sleep Wake Disorders; Smoking; Overweight; Obesity; Alzheimer Disease; Atrial Fibrillation; Heart Diseases; Cognitive Dysfunction; Ischemic Attack, Transient | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: DELPhI system — DELPhI software is acquiring and analyzing the TMS evoked response recorded with the EEG.
  Other Names: Transcranial magnetic stimulation

SUMMARY:
The DELPhi system is a software device that is used for the noninvasive evaluation of brain plasticity and connectivity. The DELPhi software uses EEG and TMS devices as accessories. Standard electro-physiological acquisition is performed using TMS to evoke regional neuronal potentials measured as EEG data. TMS-EEG data is analyzed with regards to conventional, well established characteristics of neuronal network plasticity and connectivity.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a noninvasive brain stimulation method that allows to study human cortical function in vivo. Using TMS for examining human cortical functionality is enhanced by combining TMS with simultaneous registration of electroencephalograph (EEG). EEG provides an opportunity to directly measure the cerebral response to TMS. Measuring the cortical TMS Evoked potential (TEP), is used to assess cerebral reactivity across wide areas of neocortex.

By evaluating the propagation of evoked activity in different behavioral states and in different tasks, TMS-EEG has been used to causally probe the dynamic effective connectivity of human brain networks.

In this study the sponsor is intended to collect data of subjects at the ages of 50-75, at risk for stroke and dementia using DELPHI, brain MRI scans, cognitive tests and clinical and demographic information. Some of the patients agreeing to perform a second test will serve for a reliability test.

Primary Objectives:

1. Definition of DELPHI's average TEP response of at risk for stroke and dementia population in subjects over 50-75 years old+/- STD.
2. Assessing the Safey of the use of DELPHI in at risk for stroke and dementia population.
3. Defining DELPHI's test-retest reliability by quantifying correlation coefficient between two tests.

Exploratory objectives:

1. Evaluating the sham stimulation effect.
2. Assessing confounders effecting results.

Subjects will perform a medical interview, neurological exam, cognitive evaluations, two emotional inventories and a brain MRI scan.

ELIGIBILITY:
Inclusion criteria:

1. Male and female at the ages of 50-75 years old (included) with at least one risk factor for Stroke or Dementia* and/or a suspected cognitive impairment**
2. Willing to cooperate with all study procedures. *Risk factors for Stroke and Dementia:

   * Previous stroke or TIA
   * Hypertension
   * Dyslipidemia
   * Diabetes Mellitus
   * Atrial Fibrillation
   * Other cardiac conditions (such as, MI, Valve disease etc.)
   * Smoking (any current smokers or past heavy smokers (>20 cigarettes/day)).
   * Obesity and overweight (BMI>25)
   * Familial history of dementia
   * Age ≥ 65
   * Sleep disturbances

     ** Suspected cognitive impairment:
   * self or family report of cognitive impairments
   * Objective evidence of cognitive impairments

4.2 Exclusion criteria:

1. Any neurodegenerative disease.
2. Neurological developmental disorder (e.g., Cerebral Palsy, Anoxic Brain Damage, Autism Spectrum Disorder).
3. Multiple Sclerosis (MS).
4. Major psychiatric disorders (e.g., PTSD, Bi-polar Disorder, Schizophrenia, Substance abuse),
5. Chronic pain disorders.
6. History of brain tumor, history of brain surgery or brain radiation damage.
7. Prior known epileptic episode.
8. Subjects with any metallic brain implant or fragments (such as shunt, pacemaker, clips, coils, bullet fragments, cochlear implants).
9. Subjects with any implanted devices activated or controlled by physiological signals and/or ferromagnetic or other magnetic sensitive metals implanted in the head or anywhere within 12 inches/30 cm from the stimulation coil.
10. Any contraindication to MRI.
11. With any known significant head trauma in the medical history (e.g. loss of consciousness, altered consciousness, diagnosed evidence of contusion on brain imaging following trauma.
12. Current ongoing use of opioids, anti-psychotic, or anti-epileptic medications.
13. Intake of any other CNS directed medication such as sleeping pills, SSRIs, Anxiolytics 12 hours or less prior to the DELPHI evaluation.
14. Subjects that report drug abuse.
15. Pregnant or breastfeeding woman.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: N= 300 subjects recruited by advertisements or from exsiting database at the ages of 50-75, at risk to develop stroke or dementia.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Establishing DELPhI's norms of population 50-75 years old at risk for stroke and dementia | 1 visit
  Mean, STD, standard error (SEM), coefficient of variation (CV%), minimum, median, maximum and 95% confidence interval, for every DELPHI parameter in at risk for stroke and dementia population.
Establish DELPhI's safety in subjects 50-75 at risk for stroke and dementia. | 1 week
  Rates and Frequencies of Adverse events and descriptive report of Adverse events and possible relationship to DELPHI.
DELPHI's reliability | 1 visit
  Examining DELPHI's reliability by defining Intra-Class Correlation (ICC) coefficients between two tests performed at different days and/or different operators at each of DELPHI's parameters.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Diablo Clinical Research Inc., Walnut Creek, California
  - Neurotrials Research, Atlanta, Georgia
  - Clinical Research Center CTI, Norwood, Ohio
- Sourasky Tel-Aviv Medical Center, Tel Aviv, Center, Israel

IPD SHARING:
Plan to Share IPD: No